CLINICAL TRIAL: NCT04811469
Title: A Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Study in Healthy Subjects to Evaluate the Safety, Tolerability, and Pharmacokinetics of CBP-174 After Oral Administration
Brief Title: Safety, Tolerability and Pharmacokinetics of CBP-174 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Connect Biopharma Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Organization: Connect Biopharm LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBP-174AU001
Record Dates: First submitted 2020-08-16; First posted 2021-03-23 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Healthy Adult Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBP-174 (Experimental): CBP-174 oral solution
  Interventions: Drug: CBP-174
- Placebo (Experimental): placebo oral solution
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CBP-174 — CBP-174 oral solution, given once
  Arms: CBP-174
Drug: Placebo — Placebo oral solution, given once
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of CBP-174 after a single oral dose in healthy adult subjects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single ascending dose study in healthy subjects to evaluate the safety, tolerability and pharmacokinetics of CBP-174 compared to placebo. The study plans to set 6 dose escalation cohorts with single oral dose. Each subject will receive only one dose regimen in this study and the total duration to participate the study is approximately 1 to 4-week.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled into the study only if they meet ALL of the following inclusion criteria:

1. Subjects are fully informed of the study, and are willing to participate in the study and sign the informed consent document prior to any procedure
2. Healthy male and female subjects, aged 18 to 55 years (both inclusive)
3. Body mass index is between 18 and 32 kg/m2 (both inclusive), the weight of male subjects ≥ 50 kg, the weight of female subjects ≥ 45 kg
4. Considered generally normal or abnormal with no clinical significance upon medical history, physical examination, vital signs, ECG, and clinical laboratory tests, as judged by the Investigator
5. Female subjects of child-bearing potential must agree to use highly effective contraceptive methods 1 month before the screening, during the entire study, and within 3 months after the end of this study, and have no egg donation plan within 3 months of study end. The male partner of a female subject must agree to use condoms during the screening, entire study, and within 3 months after the end of this study. Male subjects considered fertile must agree to not plan to father a child, donate sperm, and take effective contraceptive methods during the screening, entire study, and within 3 months after the end of this study. The female partner of male subjects must agree to use a highly effective method of female contraception (Section 9.8.3.2) during the screening, entire study, and within 3 months after the end of this study. Contraceptive requirements applies to subjects in same sex relationships for male and female subjects, female subjects of non child bearing potential or male subjects with female partners of non-childbearing potential.
6. Subjects who are able to communicate well with Investigators, as well as understand and adhere to the requirements of this study

Exclusion Criteria:

Subjects will be excluded from the study, if they meet ANY of the following criteria:

Subjects will be excluded from the study, if they meet ANY of the following criteria:

1. Subjects who have difficulties in venous blood collection or history of dizziness with blood or needles
2. Female subjects who have a positive pregnancy test or are breastfeeding
3. Subjects who have allergy/hypersensitivity history to any excipient of CBP-174 solution, or hypersensitivity to antihistamines, or severe allergies at the discretion of Investigator
4. Exposure to any other investigational medicinal product or any other clinical trial within 30 days or 5 times half-lives (whichever is longer) before dosing current study medication
5. Subjects who have a history of gastrointestinal (such as duodenal ulcer, alimentary tract hemorrhage, etc.), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
6. Subjects who have a history of significant eye diseases (such as keratitis, and scleritis, etc.) or clinical significant eye signs (conjunctiva hyperemia, etc.)
7. Subjects who have a history of attention deficit disorder (ADD) or attention deficit hyperactivity disorder (ADHD)
8. Subjects who have a history of sleep disorders within 2 years before the screening visit or score highly on the PSQI or ISI questionaire; or have a history of epilepsy or other seizure disorder

   *Pittsburgh Sleep Quality Index (PSQI) ≥ 8 or Insomnia Severity Index (ISI) ≥ 8
9. Subjects who have the medical history of other significant diseases (including but not limited to pulmonary, cardiovascular, gastrointestinal, hematological endocrinological, immunological, dermatological, malignant diseases, mental and nervous systems, and other related diseases) or any other disease/ailment at the discretion of the Investigator
10. Subjects with any of the following clinical laboratory tests results at screening:

    a Aspartate aminotransferase (AST) > 1.5 × the upper limit of normal (ULN)

    b Alanine aminotransferase (ALT) > 1.5 × ULN

    c Serum creatinine > 1.2 × ULN; or creatinine clearance < 60 mL/min (calculated by the Cockcroft-Gault)

    *The clinical laboratory tests of hematology, blood biochemistry, or urinalysis could be allowed repeat once if Investigator considers it necessary
11. Subjects whose QTcF interval prolongation at screening (male: QTcF interval ≥ 450 ms, female: QTcF interval ≥ 470 ms)
12. Blood donation or blood loss more than 400 mL within 3 months before the screening visit
13. Subjects with a known history of drug abuse within 2 years before the screening visit; or positive drug abuse at screening
14. Weekly alcohol consumption of more than 14 units of alcohol (1 unit of alcohol = 360 mL of beer or 45 mL of spirit with the alcohol content of 40% or 150 mL of wine) in any week within the past 3 months before the screening visit; or intake of alcohol-containing products within 48 hours before the first dose, or cannot abstain from any alcohol product during the study, or positive breath alcohol test at screening or check-in (Day -1）
15. Smoking history (> 5 cigarettes per day) within 3 months before the screening visit, or cannot abstain from any tobacco products during the study, or positive urine nicotine test before randomization
16. Excessive drinking of tea, coffee, or caffeine-containing beverage (at least 8 cups per day, 1 cup = 250 mL) any day within 3 months before screening; intake of rich caffeine- or xanthine-containing food or drinks that may produce caffeine or xanthine after being metabolized (eg, coffee, tea, chocolate, cola drinks) within 48 hours before the first dose
17. Any marketed medication (prescription and nonprescription drugs) within 14 days before the first dose or within 5 times the elimination half-life or pharmacodynamic half-life of the medication (excluding oral contraceptives and low dose paracetamol at the discretion of the Investigator, or topical ointments at the discretion of the Investigator)
18. Administration of a Coronavirus Disease 2019 (COVID-19) vaccine in the past 14 days prior to dosing
19. Use of herbal medicines, dietary supplements and vitamin within 14 days before the first dose(permissible at the discretion of the Investigator)
20. Subjects who have a major surgery within 3 months before the first dose or who plan to undergo surgery during the study
21. Positive screening test for human immunodeficiency virus (HIV) antibody, hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), or hepatitis C antibody
22. Subjects who are determined as not eligible to participate in this study by the Investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-05-14 (Actual); Study Completion 2022-05-21 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events and serious adverse events | Up to 7 days post dosing
  Adverse events will be coded according to the Medical Dictionary for Regulatory Activities (MedDRA) Dictionary.
Severity of adverse events and serious adverse events | Up to 7 days post dosing
  The investigator may use the CTCAE V5.0 to assist in the determination of severity and clinical significance.
Change in blood pressure | Up to 7 days post dosing
  Blood pressure measured in mmHg
Change in pulse rate | Up to 7 days post dosing
  Pulse rate measured per minute
Change in respiratory rate | Up to 7 days post dosing
  respiratory rate measured in breaths per minute
Change in tympanic temperature | Up to 7 days post dosing
  tympanic temperature measured in celsius
Clinically significant abnormality in physical examinations | Up to 7 days post dosing
  Physical examinations includes examination in cutaneous, lymph node, head (especially of eyes) and neck, chest, abdomen, musculoskeletal and nervous systems.
Clinically significant change in heart rate | Up to 7 days post dosing
  Heart rate in beats per minute (Bpm) through 12-lead ECG assessment. The Investigator or designee will be responsible for review and interpretation of safety ECGs on site.
Clinically significant change in RR interval | Up to 7 days post dosing
  R-R interval measured in millisecond through 12-lead ECG assessment. The Investigator or designee will be responsible for review and interpretation of safety ECGs on site.
Clinically significant change in PR interval | Up to 7 days post dosing
  P-R interval measured in millisecond through 12-lead ECG assessment. The Investigator or designee will be responsible for review and interpretation of safety ECGs on site.
Clinically significant change in QRS complex | Up to 7 days post dosing
  QRS complex measured in millisecond through 12-lead ECG assessment. The Investigator or designee will be responsible for review and interpretation of safety ECGs on site.
Clinically significant change in QT interval | Up to 7 days post dosing
  QT interval measured in millisecond through 12-lead ECG assessment. The Investigator or designee will be responsible for review and interpretation of safety ECGs on site.
Clinically significant change in Fridericia's Correction QT (QTcF) interval | Up to 7 days post dosing
  QTcF interval measured in millisecond through 12-lead ECG assessment. The Investigator or designee will be responsible for review and interpretation of safety ECGs on site.
Clinically significant abnormal laboratory value in Total Protein (TB) | Up to 7 days post dosing
  Measured in g/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Albumin (ALB) | Up to 7 days post dosing
  Measured in g/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Alanine aminotransferase (ALT) | Up to 7 days post dosing
  Measured in IU/L. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Aspartate aminotransferase (AST) | Up to 7 days post dosing
  Measured in IU/L. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Alkaline phosphatase (ALP/AKP) | Up to 7 days post dosing
  Measured in IU/L. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Glutamyl transpeptidase | Up to 7 days post dosing
  Measured in U/L. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Total bilirubin | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Direct Bilirubin | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Indirect Bilirubin | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Glucose | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Urea | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Uric Acid | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Creatinine | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Creatine Kinase | Up to 7 days post dosing
  Measured in IU/L. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Potassium | Up to 7 days post dosing
  Measured in mmol/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Sodium | Up to 7 days post dosing
  Measured in mmol/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Chloride | Up to 7 days post dosing
  Measured in mmol/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Calcium | Up to 7 days post dosing
  Measured in mmol/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Total Cholesterol | Up to 7 days post dosing
  Measured in mmol/L. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal laboratory value in Blood Triglycerides | Up to 7 days post dosing
  Measured in mmol/L. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Leukocyte Count | Up to 7 days post dosing
  Counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Neutrophil count | Up to 7 days post dosing
  Counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Lymphocyte count | Up to 7 days post dosing
  Counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Monocytes count | Up to 7 days post dosing
  Counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Eosinophils count | Up to 7 days post dosing
  Counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Basophil count | Up to 7 days post dosing
  Counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in percentage of Neutrophil | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in percentage of Lymphocyte | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in percentage of Monocytes | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in percentage of Eosinophils | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in percentage of Basophils | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Erythrocyte count | Up to 7 days post dosing
  Counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Hemoglobin | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Hematocrit | Up to 7 days post dosing
  Measured in %. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Platelets | Up to 7 days post dosing
  Counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal finding in Urine Occult Blood | Up to 7 days post dosing
  Urine Occult Blood will be record as positive or negative. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urine Bilirubin | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urine pH | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urine Protein | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urine Glucose | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urine Specific gravity | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urine Ketones | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urobilinogen | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urinary leukocyte | Up to 7 days post dosing
  Urinary leukocyte will be counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urine erythrocytes | Up to 7 days post dosing
  Urine erythrocytes will be counted in K/uL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Urine Nitrites | Up to 7 days post dosing
  Measured in mg/dL. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Prothrombin time (PT) | Up to 7 days post dosing
  Measured in seconds by coagulation tests. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Activated partial thromboplastin time (APTT) | Up to 7 days post dosing
  Measured in seconds by coagulation tests. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in International normalized ratio (INR) | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Fibrinogen (FIB) | Up to 7 days post dosing
  Measured in mmol/L. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal change in Thrombin time (TT) | Up to 7 days post dosing
  Measured in seconds by coagulation tests. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal in Feces colour | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal in Feces properties | Up to 7 days post dosing
  The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal in Fecal Red blood cell | Up to 7 days post dosing
  Measured in Units. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal in Fecal White blood cell | Up to 7 days post dosing
  Measured in Units. The physician will judge whether an abnormality is clinically significant.
Clinically significant abnormal in Fecal Occult blood | Up to 7 days post dosing
  Recorded as positive or negative. The physician will judge whether an abnormality is clinically significant.

SECONDARY OUTCOMES:
AUC0-72 h: Area under the plasma concentration-time curve of CBP-174 from time 0 to 72h | Up to 72 hours post dosing
  Calculated by non-compartmental analysis with WinNonlin (Version 8.3.1 or above)
AUC0-∞: Area under the plasma concentration-time curve of CBP-174 from time 0 to infinity | Up to 72 hours post dosing
  Calculated by non-compartmental analysis with WinNonlin (Version 8.3.1 or above)
Cmax: Maximum observed concentration | Up to 72 hours post dosing
  Calculated by non-compartmental analysis with WinNonlin (Version 8.3.1 or above)
Tmax: Time to maximum concentration; | Up to 72 hours post dosing
  Calculated by non-compartmental analysis with WinNonlin (Version 8.3.1 or above)
T1/2: Elimination half-life; | Up to 72 hours post dosing
  Calculated by non-compartmental analysis with WinNonlin (Version 8.3.1 or above)
λz: Terminal phase rate constant; | Up to 72 hours post dosing
  Calculated by non-compartmental analysis with WinNonlin (Version 8.3.1 or above)
CL/F: Apparent clearance; | Up to 72 hours post dosing
  Calculated by non-compartmental analysis with WinNonlin (Version 8.3.1 or above)
V/F: Apparent Volume; | Up to 72 hours post dosing
  Calculated by non-compartmental analysis with WinNonlin (Version 8.3.1 or above)
%AUCex: Percentage of AUC0-∞ obtained by extrapolation | Up to 72 hours post dosing
  Calculated by non-compartmental analysis with WinNonlin (Version 8.3.1 or above)

CONTACTS AND LOCATIONS:
Overall Officials: Australia Connect, Study Director — Connect Biopharma Australia Pty Ltd; Suzhou Connect, Study Director — Connect Biopharm LLC
Locations (1):
- Nucleus Network Pty Ltd, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No